CLINICAL TRIAL: NCT04418960
Title: Physiological Changes of the Mitral Annulus After Annuloplasty in Barlow Disease: an MRI-focused Study
Brief Title: Physiological Changes of the Mitral Annulus After Annuloplasty in Barlow Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-02240; ch20Grapow
Record Dates: First submitted 2020-05-12; First posted 2020-06-05 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Barlow Disease (BD); Mitral Insufficiency
Keywords: mitral annuloplasty; mitral valve repair; mitral annulus; coaptation of mitral leaflets
MeSH Terms: conditions — Mitral Valve Insufficiency | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Magnetic resonance imaging (MRI) — MRI pre- and postoperatively for detailed analysis of the ventricle and the mitral annulus. The first MRI will be performed on the admission day before surgery. The second MRI will be performed during the hospital stay, between 3 and 7 days after the operation. The MRI images are interpreted through a specialized cardiologist and radiologist.

SUMMARY:
Barlow disease (BD) is a common cause of mitral insufficiency. In 2012 the University Hospital of Basel started to perform a simplified mitral valve repair technique in BD just by implanting an annuloplasty-ring. It is hypothesized that the major mechanism of the valvular insufficiency in Barlow disease is a deformation of the left ventricle and the posterior mitral annulus, causing its aberrant displacement during the systole towards posterior and basal and thus impairing the coaptation of the leaflets. This prospective individual MRI study is to investigate the ventricle and the mitral annulus pre- and postoperatively for detailed analysis.

ELIGIBILITY:
Inclusion Criteria:

* identified Barlow disease suffering from significant mitral insufficiency with indication to surgery

Exclusion Criteria:

* Active endocarditis or any other etiology of mitral insufficiency else than Barlow disease
* Inability to perform a cardiac MRI (e.g., metallic implants, claustrophobia)
* Pregnancy
* Inability to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to cardiac surgery clinic (University Hospital Basel) through cardiologist meeting the inclusion criteria based on the medical history, clinical and echocardiographic findings.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2018-09-21 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Change in anatomical structures by MRI | The first MRI will be performed on the admission day before surgery. The second MRI will be performed during the hospital stay, between 3 and 7 days after the operation.
  Change in anatomical structures by MRI: distance (mm) between the mitral annulus and the cardiac apex during the cardiac cycle before and after surgical correction

SECONDARY OUTCOMES:
function of the mitral valve by echocardiography | during the hospital stay, between 3 and 7 days after the operation and at cardiological follow-up over the first 3 months.
  association between reduction of movement of the posterior annulus and the function of the valve after surgery (i.e. its residual insufficiency (0 = absent, 1 = mild, 2 = moderate, 3 = severe)). Evaluated with echocardiography as it is routinely performed in cardiac surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Grapow, Prof. Dr. med., Principal Investigator — HerzZentrum Hirslanden, Zurich
Locations (1):
- Cardiac Surgery, University Hospital Basel, Basel, Switzerland